CLINICAL TRIAL: NCT03796949
Title: Threatened Preterm Birth and Time of Subsequent Delivery; Prediction Model Based on Biomarkers and Maternal/Obstetrical Characteristics
Brief Title: Threatened Preterm Birth and Time of Subsequent Delivery -a Prediction Model
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Marie Blomberg, Professor, Linkoeping University
Other Study IDs: 960624abc
Record Dates: First submitted 2019-01-07; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Preterm Birth; Immunologic Activity Alteration
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples Serum samples RNA samples Placental biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- threatened preterm birth: Women with either preterm labor or preterm prelabor rupture of the membranes. Blood samples taken at time of inclusion in the study.
- Controls: Women with normal pregnancies. Blood samples taken at time of inclusion in the study, either prelabor (during pregnancy) or during active phase of labor.

SUMMARY:
This study investigates immunological and clinical markers in threatened preterm birth aiming to create a prediction model for preterm birth.

DETAILED DESCRIPTION:
Preterm birth is the main cause of neonatal mortality and morbidity and despite a lot of effort the mechanisms leading to preterm birth are poorly understood. In threatened preterm birth it is difficult to identify the true high risk cases ultimately leading to preterm birth. These women are often overtreated.

In this study blood samples are taken from women with threatened preterm birth and from women with normal pregnancies before and during labor.

Differences in clinical characteristics and immunological markers between the groups are studied in order to design a prediction model for preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* Threatened preterm birth before 34 weeks of gestation; either threatened preterm labor and/or preterm prelabor rupture of the membranes
* Age > 18 years
* Swedish-speaking (understanding study information)

Exclusion Criteria:

* Multiple gestation
* Blood borne infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 women with threatened preterm labor before 34 weeks of gestation, 40 women with preterm prelabor rupture of the membranes before 34 weeks of gestation, 40 women with normal pregnancies in labor at term, 44 women with normal pregnancies during pregnancy (before labor)
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Time of delivery | Outcome noted at delivery
  Delivery before 34 weeks of gestation or after 34 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Marie Blomberg, MD PhD, Principal Investigator — Department of Obstetrics and Gynecology, Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No